CLINICAL TRIAL: NCT02737631
Title: Human Repeat Insult Patch Test to Evaluate Personal Lubricants
Acronym: HRIPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Church & Dwight Company, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ST-7619
Record Dates: First submitted 2016-02-29; First posted 2016-04-14 (Estimated); Results first posted 2017-09-01 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-03

CONDITIONS: Erythema; Edema
MeSH Terms: conditions — Erythema; Edema

STUDY DESIGN:
Masking Description: All participants receive the same interventions

ARMS (1):
- Healthy subject (Experimental): Healthy subjects exposed to "Chameleon" personal lubricant via occlusive patch
  Interventions: Device: "Chameleon" Personal Lubricant

INTERVENTIONS:
Device: "Chameleon" Personal Lubricant

SUMMARY:
The purpose of this test is to evaluate the sensitizing potential of a personal lubricant, as a result of repeated occlusive patch. The intervention will be applied for a total of 9 induction applications, followed by an approximately 2 week rest period, then followed by a 24-72 hour Challenge applications.

ELIGIBILITY:
Inclusion Criteria:

* good health as determined from screener
* signed and dated informed consent
* signed and dated HIPAA Form

Exclusion Criteria:

* subjects on test at any other research laboratory or clinic
* known allergy or sensitivity to cosmetics and toiletries, including sunscreens, adhesives and/or topical drugs
* pre-existing dermatologic conditions which have been diagnosed by a medical professional (e.g. psoriasis, eczema, etc.) which would interfere with this study
* pre-existing other medical conditions (e.g. adult asthma, diabetes).
* treatment with antibiotics, antihistamines or corticosteroids within two weeks prior to initiation of the test
* chronic medication which could affect the results of the study (e.g., insulin, corticosteroids, antihistimines, steroidal or non-steroidal anti-inflammatory drugs [except for therapeutic maintenance dosage of aspirin], antibiotics, steroid inhalers, etc.)
* known pregnant or nursing women

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2016-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynne B Harrison, PhD, Principal Investigator — Harrison Research Laboratories, Inc.
Locations (1):
- Harrison Research Laboratories, Inc., Union, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Subject: Healthy subjects exposed to Trojan "Chameleon" personal lubricant via occlusive patch
  Trojan "Chameleon" Personal Lubricant
Period: Overall Study
Arm/Group | Healthy Subject
Started | 222
Completed | 222
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Subject
Number analyzed (Participants) | 222
Age, Customized [Count of Participants; unit: Participants]
  18-69 years | 222
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150
  Male | 72
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients That Showed Sensitization Reaction to the Test Material at Challenge
Time Frame: 24, 48 and 72 hours after patch application
Measure: Count of Participants; unit: Participants
Groups:
- Healthy Subject: Healthy subjects exposed to "Chameleon" personal lubricant via occlusive patch
  "Chameleon" Personal Lubricant
Arm/Group | Healthy Subject
Number analyzed (Participants) | 222
Participants | 0

ADVERSE EVENTS:
Arm/Group | Healthy Subject
Serious Adverse Events (participants affected / at risk) | 0/222
Other Adverse Events (participants affected / at risk) | 0/222

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Confidentiality agreement in place with PIs.